CLINICAL TRIAL: NCT07179939
Title: A Multicenter, Open-Label, Phase II Trial of Exploring the Maintenance of Trastuzumab Plus Pyrotinib or Trastuzumab Plus Dalpiciclib and Endocrine Therapy Based on HR Status Following Trastuzumab Rezetecan as Induction Treatment for HER2 Positive Unresectable Locally Recurrent or Metastatic Breast Cancer
Brief Title: Maintenance Therapy in HER2-Positive Unresectable Locally Recurrent or Metastatic Breast Cancer: A Phase II Study
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry); Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-BC-II-111
Record Dates: First submitted 2025-08-06; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-08

CONDITIONS: HER2-positive Breast Cancer
MeSH Terms: interventions — pyrotinib; dalpiciclib; Trastuzumab; Anastrozole; exemestane; Fulvestrant; Leuprolide; Goserelin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Experimental (Experimental): All patients will receive a 6-cycle induction phase with T-DXh 4.8 mg/kg body weight administered as an intravenous (IV) infusion on day 1 (D1) of each 21-day cycle (Q3W).
  Participants may continue with maintenance treatment if T-DXh is discontinued prematurely due to unacceptable toxicity prior to disease progression.
  During the maintenance phase, participants with HR positive disease will receive trastuzumab combined with dalpiciclib and endocrine therapy and for those with HR negative disease will receive trastuzumab combined with pyrotinib.
  Interventions: Drug: Trastuzumab rezetecan; Drug: Pyrotinib; Drug: Dalpiciclib; Drug: Trastuzumab; Drug: ET: Letrozole/ Anastrozole/ Exemestane/ Fulvestrant/ Leuprorelin/ Goserelin.

INTERVENTIONS:
Drug: Trastuzumab rezetecan — Trastuzumab rezetecan is a lyophilized powder for injection intravenously. Administered according to label.
  Other Names: SHR-A1811; T-DXh
Drug: Pyrotinib — 320 mg/d, q.d., p.o. A course of treatment need 21 days.
Drug: Dalpiciclib — 125 mg/d, q.d., p.o. day 1-21, every 28 days.
Drug: Trastuzumab — Administered according to label.
Drug: ET: Letrozole/ Anastrozole/ Exemestane/ Fulvestrant/ Leuprorelin/ Goserelin. — Administered according to label.

SUMMARY:
This is a phase II trial exploring the maintenance therapy with trastuzumab combined with pyrotinib or dalpiciclib and endocrine therapy in HER2-positive advanced breast cancer based on different hormone receptor (HR) statuses following trastuzumab rezetecan (T-DXh, SHR-A1811) as induction treatment for HER2-positive unresectable locally recurrent or metastatic breast cancer (MBC) patients.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this trial, an individual must meet ALL the following criteria:

1. Patient must be capable to understand the purpose of the study and have signed written informed consent form (ICF) prior to beginning specific protocol procedures.
2. Female patients ≥ 18 years of age at the time of signing ICF.
3. Breast Cancer Requirements:

   1. Histologically or cytologically confirmed HER2-positive(IHC 3+ or ISH+) unresectable locally advanced or metastatic breast cancer (Note: Patients eligible for curative-intent treatment are excluded).
   2. Documented hormone receptor (HR) status.
   3. No prior systemic anti-tumor therapy for recurrent/metastatic disease (≤1 line of endocrine therapy is permitted*).
   4. For patients who received (neo)adjuvant therapy: >12 months between the end of systemic treatment (excluding endocrine therapy) and recurrence/metastasis.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
5. Adequate Organ Function.
6. Pregnancy and Contraception: Women of childbearing potential (WOCBP) must agree to use highly effective contraception from screening until7 months after the last dose of study treatment and must refrain from breastfeeding.

Exclusion Criteria:

An individual who meets ANY of the following criteria will be excluded from participation in this trial:

1. Known active CNS metastases not treated with surgery or radiotherapy, except for those who have achieved stable disease for ≥1 month after treatment and have discontinued corticosteroids for >2 weeks.
2. Received major cancer-related surgery, radiotherapy, chemotherapy, immunotherapy, molecular targeted therapy, biologic therapy, or investigational drug therapy within 4 weeks prior to the first dose of study treatment.
3. Previous treatment with antibody-drug conjugates containing exatecan derivative topoisomerase I inhibitors.
4. Presence of clinically significant cardiovascular conditions, including:

   1. Severe/unstable angina
   2. Symptomatic congestive heart failure (NYHA class ≥II)
   3. Clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention
   4. Myocardial infarction within 6 months before the first dose
5. Has a history of non-infectious interstitial lung disease (ILD)/pneumonitis that required steroids, has current ILD/pneumonitis, or has suspected ILD/pneumonitis that cannot be ruled out by imaging at screening.
6. Known substance abuse or any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, contraindicate patient participation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2025-09-10 (Estimated); Primary Completion 2030-12-30 (Estimated); Study Completion 2031-12-30 (Estimated)

PRIMARY OUTCOMES:
PFS | From the date of treatment initiation until to the first occurrence of disease progression as determined locally by the investigator assessment using RECIST v.1.1 or death from any cause, whichever occurs first，assessed up to 60 months
  Defined as the period from treatment initiation until to the first occurrence of disease progression as determined locally by the investigator assessment using RECIST v.1.1 or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
OS | From the date of treatment initiation to the death from any cause, assessed up to 84 months
  Defined as the period from treatment initiation to death from any cause, as determined locally by the investigator.
Objective response rate (ORR) | At least 4 weeks after first documented response
  Defined as the rate of patients with complete response (CR) or partial response (PR), as determined locally by the investigator using RECIST v.1.1.
Safety and tolerability | From the date of treatment initiation until to the discontinuation of treatment，assessed up to 60 months
  Assessed in all patients as per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University, Shanghai, China